CLINICAL TRIAL: NCT07223554
Title: A Tailored, Web-Based Self-Management Program to Treat Pain in Chronic Pancreatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jorge Machicado, MD, MPH, Clinical Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00277458
Record Dates: First submitted 2025-10-29; First posted 2025-11-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pancreatitis
Keywords: Behavioral intervention; Self-management; Pain
MeSH Terms: conditions — Pancreatitis, Chronic; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-based self-management program (Experimental): Participants will be assigned to a web-based, self-management program that has been adapted to chronic pancreatitis. Participants will participate in this program for 12 weeks.
  Interventions: Behavioral: Web-based self--management program

INTERVENTIONS:
Behavioral: Web-based self--management program — Participants in this study will be granted access to the adapted website after participants complete baseline questionnaires. All participants will be encouraged to engage with all the sections of the website. From week 1 to 4, participants will receive a single standardized guidance to complete one module a week on generic pain modules. From weeks 5 to 12, participants will receive weekly tailored messaging that will direct participants to specific modules based on individual survey scores from the baseline assessments.

SUMMARY:
This research study aims to evaluate the feasibility and acceptability of a web-based, self-guided, disease-specific self-management program tailored to individual health status profiles for patients with painful chronic pancreatitis.

DETAILED DESCRIPTION:
This is a single center, prospective, open-label, pilot trial of 30 patients with painful chronic pancreatitis (CP). Participants will be assigned to a 12-week web-based, self-management program known as PainGuide that has been adapted to CP. Participants will receive specific instruction to complete one module a week over the first 4 weeks. Next, participants will receive weekly tailored messaging for the last 8 weeks using symptom scores from baseline assessments and will be asked to complete modules that best address participants symptoms. Participants will complete online surveys at baseline, 4 weeks, 8 weeks, and 12 weeks, and will be interviewed at the end of program to understand participants perceptions on the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of chronic pancreatitis.
* Abdominal pain for ≥ 3 months and of intensity rated at least 4 or higher on a 0-10 Numeric Rating Scale at least once in the last month.
* Access to an Internet-connected device (e.g. computer or phone).

Exclusion Criteria:

* Unable to speak or read English as the web-based program is currently in English language only.
* Incarcerated individuals.
* Currently receiving chemotherapy.
* Suspected or diagnosed pancreatic cancer.
* Currently receiving psychotherapy or cognitive behavioral therapy.
* Serious visual difficulties that would limit completing the web-based program.
* Substantial cognitive impairment or mental illness that would prevent providing informed consent and completion of questionnaires.
* Any other condition, which in the opinion of the investigator would impede compliance or hinder the completion of the study.
* Actively enrolled in another clinical trial for chronic pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of enrolled participants that log in at least once during weeks 1-4 and at least once to the recommended modules during weeks 5-12. | 12 weeks
  This number is used to determine adherence to the intervention.
Proportion of participants with an average item score of ≥4 out of 5 on the Acceptability of Healthcare Interventions Questionnaire | 12 weeks
  This is a validated 8-item questionnaire that assesses acceptability using a 5-point Likert scale rated 1-5.

SECONDARY OUTCOMES:
Proportion of participants approached that enroll in the study. | Approximately 1 year (during recruitment period)
  This number is used to determine enrollment feasibility to the web-based program in patients with painful CP.
Proportion of enrolled participants that log in at least once during the 12-week program | 12 weeks
  This number is used to determine minimal adherence to the web-based program in patients with painful CP.
Proportion of enrolled participants that log in at least once a week during weeks 1-4 and at least once a week to the recommended modules during weeks 5-12. | 12 weeks
  This number is used to determine maximal adherence to the web-based program in patients with painful CP.
Number of logins per participant during the 12-week intervention | 12 weeks
  This number is used to determine engagement with the web-based program in patients with painful CP.
Proportion of fully completed questionnaires by the total number given to participants | 12 weeks
  This number is used to assess the feasibility of data collection procedures.
Proportion of participants who scores the general acceptability item on the acceptability scale ≥4 out of 5 | 12 weeks
  This is a validated 8-item questionnaire that assesses acceptability using a 5-point Likert scale rated 1-5.
Proportion of participants that feel the web-based program is easy and intuitive to use based on a usability score > 68 on the System Usability Scale (SUS) | 12 weeks
  This is a validated 10-item questionnaire that measures the perceived usability of a system focusing on ease of use, efficiency, and overall satisfaction. Participants score from 1 (strongly disagree) to 5 (strongly agree). To calculate the SUS score, respondents' ratings are adjusted: subtract 1 from the score for odd-numbered items and subtract each score from 5 for even-numbered items. The adjusted scores are then summed and multiplied by 2.5, yielding a total score ranging from 0 to 100. Generally, a SUS score above 68 indicates above-average usability, though this benchmark can vary with different systems.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Machicado, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No